CLINICAL TRIAL: NCT03025425
Title: Palliation of Dyspnea With Mouth Piece Ventilation in Acute Exacerbation of COPD Without Respiratory Insufficiency
Brief Title: Palliation of Dyspnea With Mouth Piece Ventilation in AECOPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in finding suitable patients
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Lauri Lehtimäki, Associate Professor, Tampere University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R16148_TAYS
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: COPD Exacerbation; Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MPV-arm (Experimental): Subjects use mouth piece ventilation (MPV) according to their will for 24 hours to alleviate dyspnea.
  Interventions: Device: Trilogy 100 ® (Philips Respironics)

INTERVENTIONS:
Device: Trilogy 100 ® (Philips Respironics) — Mouth piece Ventilation (MPV) using Trilogy 100 ® (Philips Respironics).

SUMMARY:
An uncontrolled feasibility study on using mouth piece ventilation in palliation of dyspnea in subjects with acute exacerbation of COPD without acute hypercapnic respiratory failure. Subjects are recruited from the local respiratory ward. The main outcomes are the compliance of the subjects with the treatment and alleviation of dyspnea during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* a previous diagnosis of COPD
* hospitalized due to acute exacerbation of COPD
* at least moderate dyspnea (NRS = Numeric Rating Scale ≥ 4)
* no acute hypoventilation (pH ≥ 7.35 and PCO2 ≤ 6.0 kPa)
* able to understand the study and to give informed consent

Exclusion Criteria:

* unable to participate and use MPV due to e.g. delirium or lack of co-operation
* acute hypoventilation (pH < 7.35 or PCO2 > 6.0 kPa)
* acute need for ventilatory support
* the cause of the dyspnea can be successfully treated
* unable to give informed consent
* a previous chronic hypoxemic or hypercapnic respiratory insufficiency that has been treated on a long-term basis also at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Change in dyspnea after initial period of using MPV | 5-60 min
  Change in dyspnea after initial period of using MPV

SECONDARY OUTCOMES:
Change in dyspnea after 24 hours of using MPV | 24 hours
  Change in dyspnea after 24 hours of using MPV
Proportion of subjects having side-effects or not being compliant with MPV | 24 hours
  Proportion of subjects having side-effects or not being compliant with MPV
Proportion of subjects gaining from MPV | 24 hours
  Proportion of subjects gaining from MPV
Proportion of subjects willing to continue on MPV after the intervention | 24 hours
  Proportion of subjects willing to continue on MPV after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Lehtimäki, MD, Principal Investigator — Tampere University Hospital, Allergy centre
Locations (1):
- Dpt of Respiratory Medicine, Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Derived] Leivo-Korpela S, Rantala HA, Piili RP, Lehtimaki L, Lehto JT. Palliation of Dyspnea With Mouthpiece Ventilation in Patients With Chronic Obstructive Pulmonary Disease: A Pilot Feasibility Study. J Palliat Med. 2023 Sep;26(9):1261-1265. doi: 10.1089/jpm.2023.0039. Epub 2023 May 4. PMID 37155710